CLINICAL TRIAL: NCT04838236
Title: Improving Access to Cigarette Cessation Treatment Among African American Smokers: Development and Evaluation of an Integrated mHealth Application
Brief Title: Smoking, Stress, and Mobile Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Houston (Other)
Collaborators: University of Oklahoma (Other)
Responsible Party: Principal Investigator, Michael J. Zvolensky, Ph.D., Hugh Roy and Lillie Cranz Cullen Distinguished University Professor, University of Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000360
Record Dates: First submitted 2021-03-25; First posted 2021-04-09 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Smoking, Tobacco
MeSH Terms: conditions — Tobacco Smoking | interventions — Nicotine Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MASP app + NRT (Experimental): MASP is an intervention designed to assist African American smokers with anxiety sensitivity quit smoking through the use of educational videos, tailored messages, and interoceptive exercises designed to help the user overcome negative feelings of stress and nicotine withdrawal.
  Interventions: Other: MASP app + NRT
- QuitGuide app + NRT (Other): The QuitGuide app is a standard of care app that allows users to track their nicotine cravings, and provides users with motivational messages.
  Interventions: Other: QuitGuide app + NRT

INTERVENTIONS:
Other: MASP app + NRT — MASP is a mobile intervention that targets anxiety sensitivity among African American smokers (Mobile Anxiety Sensitivity Program for Smoking: MASP). Our intervention is framed within the cultural context of interoceptive stress among African American smokers, which is supported by theory, empirical evidence, and characteristics of this group. The MASP app employs a variety of features to educate its users on how to deal with stress, anxiety, and nicotine withdrawal symptoms. The app contains a series of on-demand features, including a coping toolkit, stress management trainings, and a series of educational videos. MASP also utilizes Ecological Momentary Assessments (EMAs) to gather information, and provide personalized messages to users in real time.
  Arms: MASP app + NRT
Other: QuitGuide app + NRT — Quitguide is a smartphone-based National Cancer Institute (NCI) app for standard mobile smoking cessation treatment. The app contains features that allows its' users to better understand their smoking patters, and build skills needed to becomes and stay smoke free. The app allows users to track their cravings, and delivers motivational messages to users for each craving they track.
  Arms: QuitGuide app + NRT

SUMMARY:
We seek to refine and evaluate the novel mobile intervention, Mobile Anxiety Sensitivity Program for Smoking (MASP) which was initially developed and previously tested by our team, targeting sensitivity to interoceptive stress, and to apply it among African American smokers. Our culturally adapted intervention is framed within a sociocultural context of interoceptive stress, which is supported by theory, empirical evidence, and characteristics of African American smokers. The MASP app contains educational content on the history of tobacco and the African American community.

DETAILED DESCRIPTION:
The objective of the current trial is to refine and conduct a comprehensive cultural adaptation of an initially tested novel, mobile intervention that targets anxiety sensitivity (AS) among African American smokers (MASP). The MASP app checks in with users throughout the day to assess their mood, whether or not they're experiencing any cravings or withdrawal symptoms, and their overall mental health. When users indicate they are struggling with staying abstinent, or if they are experiencing heighted levels of stress or anxiety, the app selects and delivers a tailored message from its library of hundreds of messages and videos. For instance, if a user indicates they are struggling with nicotine cravings, and feel as though they are about to smoke, they will receive an individually tailored suggestion on how to cope with the feeling, and strategies to act and overcome it. The app also contains videos that are designed to teach relaxation techniques, as well as training exercises that teach participants how to cope with uncomfortable feelings of stress and nicotine withdrawal they are likely to experience while quitting nicotine. The MASP app has the potential to deliver highly effective and accessible treatment to individuals who are looking to take that major step in their life, and quit smoking for good.

Individuals interested in participating in the study will complete informed consent and a study screener via RedCap and phone call with study staff (signatures will be obtained digitally via RedCap). Those found eligible during the phone screener will download the Insight app onto their personal phone to confirm compatibility and complete the baseline assessment. Those who do not possess a phone that is compatible with the Insight platform will be mailed a compatible phone so they can complete the baseline assessment. Upon completion of the baseline survey, participants will be mailed a Bedfont Carbon Monoxide monitor (iCO) that can be used to remotely verify smoking status, a Greenphire Mastercard, and 4 weeks of NRT. Upon receipt of the iCO, participants will complete a brief phone call to walk them through the use of the iCO and study app. Participants (N=25) in phase II will be in the study for a total of 6 weeks. Upon completion of Phase II, we will analyze data and utilize feedback collected from phase II participants to create MASP 3.0. We will then begin phase III of the study. Participants (N=220) in the study will receive either the MASP 3.0 or QuitGuide plus EMA app following the completion of the baseline assessment. Specifically, following completion on the baseline assessment they will receive a unique code that they will type into the app to place them in the group that they were randomized to. All participants will complete app-based follow-up assessments 1, 2 (quit day), 3, 4, 5, 6, 28, and 54 weeks after the baseline visit. We expect phase III of the study will be completed within a period of 30-36 months.

ELIGIBILITY:
Inclusion Criteria:

18 years of age or older, self-identify as African American, high anxiety sensitivity defined as a SSASI score of ≥ 5 assessed during phone intake via the SSASI measure (cut-off score to identify high AS individuals), daily smoking (minimum of 5 cigarettes per day) for > 2 years (assessed at pre-screening level [i.e. "Do you currently smoke cigarettes?", "How many cigarettes do you usually smoke on an average day?", "How long have you been smoking at that rate?"] and screening level by providing a picture of their pack of cigarettes, or ashtray in real-time to screen out non-smokers), motivated to quit smoking (≥ 5 on a 10-point scale), willing and able to complete all study surveys/assessments, willing to use NRT, and willing to quit smoking 2 weeks after completion of the baseline survey and receipt of study materials (e.g., iCO, nicotine replacement medications), reside in the United States (assessed at screening level by providing a picture of a valid United States ID card), willing to download and leave the app on the phone for the next year, is able to provide a 12-hour window within a standard day for their wake time, provide their social security number, residency status, and date of birth, Score ≥ 4 on the REALM-SF indicating > 6th grade English literacy level (needed to complete EMAs).

Exclusion Criteria:

Report of current or intended participation in a concurrent substance abuse treatment, ongoing psychotherapy of any duration directed specifically toward the treatment of anxiety or depression, not being fluent in English, current use of any pharmacotherapy or psychotherapy for smoking cessation not provided by the researchers (via self-report during the phone screen), legal status that will interfere with participation (provided via self-report during the phone screen), cognitive impairment (assessed via the 6-item Cognitive Impairment Test (6CIT)), non-African American, younger than 18, high blood pressure that is not under control, has experienced a heart attack (myocardial infarction) within the past 2 weeks, pregnant or breastfeeding, or planning to become pregnant within the next 6 months. Those who participated in a previous stage of the study will not be eligible to participate in further study stages. Individuals who identify themselves as undocumented immigrants will not be eligible to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2021-12-20 (Actual); Primary Completion 2025-04-25 (Actual); Study Completion 2025-04-25 (Actual)

PRIMARY OUTCOMES:
A qualitative interview will be used to evaluate the mobile app for style and presentation, perceived utility, ease of use, usefulness of features, and willingness to refer to a friend. | Week 6 follow-up (Phases II and III)
  the Qualitative Interview is a 21-item interview that aims to assess participant experiences with the smartphone applications. This interview will be conducted at the 6-week follow-up phone interview (end-of-treatment) and will be recorded for qualitative data analysis. Patient adherence will be assessed through examination of treatment components that are used within each app (e.g., videos watched, compliance with homework and exposure exercises with a standardized rating scale).
Levels of satisfaction and perceived treatment quality regarding the intervention, as assessed by the Treatment Quality and Satisfaction Survey | Week 6 follow-up (Phases II and III)
  The Treatment Quality and Satisfaction Survey was developed for the purposes of this study. This 22-item measure assesses participants' experiences during the treatment period and while using the smart phone application.
Change in Carbon Monoxide levels at Baseline as measured by the Carbon Monoxide Analysis (Phone Bedfont iCO Smokerlyzer) at follow up appointments. | From Baseline to end of study (Phase II end of study = Week 6 follow up; Phase III end of study = 54 week follow up)
  Our primary study outcome will be biochemically confirmed 7-day point prevalence abstinence. The Bedfont iCO Smokerlyzer will be used to verify smoking status during the follow-up assessments. The monitors attach to the smartphone and will be used to remotely verify self-reported smoking abstinence during phone-based monitoring periods over the post-quit period. Our CO criteria for abstinence is consistent with numerous studies using cutoffs of < 7 ppm. This will be used to verify smoking status, as well as change in smoking behaviors throughout the study.

SECONDARY OUTCOMES:
Stage of ethnic identity attitudes expressed by participants as measured by the Black Racial Identity Attitude Scale | Baseline
  The Black Racial Identity Attitude Scale a 12-item scale that aims to identify the stage of racial identity development a person is in. It consists of 3 subparts: Immersion/Emersion, Pre-encounter, and Encounter. Higher scores indicate more agreement with the items. The Black Racial Identity Attitude Scale will be utilized to explore whether perceived ethnic identity functions as a moderator of smoking outcomes.
Change from Baseline in depression related impairment on the 5-item Overall Depression Severity and Impairment Scale at subsequent follow-up appointments. | From Baseline to end of study (Phase II end of study = Week 6 follow up; Phase III end of study = 54 week follow up)
  The Overall Depression Severity and Impairment Scale is a brief, five-item measure for assessing the frequency and intensity of depressive symptoms, as well as functional impairments related to depressive symptoms. Higher scores indicate higher levels of impairment related to depression symptoms. This scale will be used to evaluate the mechanisms underlying intervention effects, including depression symptoms, and the indirect effects of the intervention on smoking cessation via this mechanism of change.
Change from Baseline in anxiety related impairment on the 5-item Overall Anxiety Severity and Impairment Scale at follow-up appointments. | From Baseline to end of study (Phase II end of study = Week 6 follow up; Phase III end of study = 54 week follow up)
  The Overall Anxiety Severity and Impairment Scale is a brief continuous measure of overall anxiety severity and impairment. Higher scores indicate higher impairment as a result of anxiety. It will be used to evaluate the mechanisms underlying intervention effects, including anxiety symptoms, and the indirect effects of the intervention on smoking cessation via this mechanism of change.
Levels of acculturation expressed by participants as measured by the African American Acculturation Scale. | Baseline
  The African American Acculturation scale is a 10-item scale that assesses cultural and media preferences, racial balance, and contexts of social interaction, and race-related attitudes and comfort with Whites versus Blacks. Lower scores represent higher levels of acculturation towards the dominant culture.
Items assessing stress levels related to the COVID-19 pandemic will be utilized to explore whether COVID-19 associated stress functions as a moderator of smoking outcomes. | Baseline
  Items will assess whether participants have received testing for the corona virus, whether they have been hospitalized because of COVID, and the severity of any symptoms they have experienced. Additionally, items will also assess fears and anxieties related to the COVID-19 pandemic. Higher scores for both of these scales indicate greater stress due to the COVID-19 pandemic.
Change from week 1 follow up in withdrawal symptoms as assessed by the Minnesota Nicotine Withdrawal Scale at subsequent follow up appointments. | From Baseline to end of study (Phase II end of study = Week 6 follow up; Phase III end of study = 54 week follow up)
  The Minnesota Nicotine Withdrawal Scale is a 10-item scale used to assess severity of nicotine withdrawal symptoms. Higher scores indicate levels of nicotine withdrawal. It will be used to evaluate the mechanisms underlying intervention effects, including nicotine withdrawal, and the indirect effects of the MASP intervention on smoking cessation via this mechanism of change.
Change from Screener in levels of anxiety sensitivity on the 5-point Short Scale Anxiety Sensitivity Index at follow up appointments. | From Baseline to end of study (Phase II end of study = Week 6 follow up; Phase III end of study = 54 week follow up)
  The Short Scale Anxiety Sensitivity Index utilizes a 5-item Likert scale to measure anxiety sensitivity. Higher score indicate higher levels of anxiety sensitivity. This index will be used to evaluate the mechanisms underlying intervention effects, including the intervention effect on reductions in anxiety sensitivity, and the indirect effects of the intervention on smoking cessation via this mechanism of change.
Change in discrimination burden using the section of the Jackson Heart Study Discrimination Instrument will be used to assess whether our intervention has underlying effects on stress-based burden from racial/ethnic discrimination. | From Baseline to end of study (Phase II end of study = Week 6 follow up; Phase III end of study = 54 week follow up)
  This measure contains 4-items that assess perceptions of discrimination. Higher scores indicate higher difficulty living a productive and full life because of perceived experience of discrimination. The measure will be used to assess change in stressed based burden from racial discrimination.
Levels of perceived discrimination as measured by the Everyday Discrimination Scale. | Baseline
  The Everyday Discrimination Scale assesses perceptions of discrimination or unfair treatment. Higher scores indicate higher perceived discrimination. The Everyday Discrimination Scale will be utilized to explore whether perceived racial discrimination functions as a moderator of smoking outcomes.
Time to first lapse | From Baseline to end of study (Phase II end of study = Week 6 follow up; Phase III end of study = 54 week follow up)
  Time to first will be measured via EMAs. Participants will press a button in the app (i.e. I Already Slipped), and once this is done, MASP will record the time and date the participant reported lapsing.
Longest time of quit | From Baseline to end of study (Phase II end of study = Week 6 follow up; Phase III end of study = 54 week follow up)
  Longest time of quit will be measured via EMAs. Participants will press a button in the app (i.e. I Already Slipped), and once this is done, MASP will record the time and date the participant reported lapsing.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - TSET Health Promotion Research Center, Oklahoma City, Oklahoma
  - RESTORE Laboratory: Research on Emotion, Substance Treatment Outcomes, and Racial Equity, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cheney MK, Alexander AC, Garey L, Gallagher MW, Hebert ET, Vujanovic AA, Kezbers KM, Matoska CT, Zvolensky MJ, Businelle MS. Adapting a Mobile Health App for Smoking Cessation in Black Adults With Anxiety Through an Analysis of the Mobile Anxiety Sensitivity Program Proof-of-Concept Trial: Qualitative Study. JMIR Form Res. 2025 Feb 7;9:e53566. doi: 10.2196/53566. PMID 39918847
- [Derived] Businelle MS, Garey L, Gallagher MW, Hebert ET, Vujanovic A, Alexander A, Kezbers K, Matoska C, Robison J, Montgomery A, Zvolensky MJ. An Integrated mHealth App for Smoking Cessation in Black Smokers With Anxiety: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2022 May 30;11(5):e38905. doi: 10.2196/38905. PMID 35635746